CLINICAL TRIAL: NCT06712979
Title: Comparison Between Lee- Silverman Method and Lung Volume Recruitment Tecnhique in Voice Professionals
Brief Title: Addiction of Lung Volume Recruitment Technique in Lee Silverman Protocol for Voice Professionals
Acronym: LVRTVOICE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Ciencias da Saude (Other)
Responsible Party: Principal Investigator, Vinicius Zacarias Maldaner da silva, Mentor in Human Movement and Rehabilitation, Escola Superior de Ciencias da Saude
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LVRT VOICE TRAINING
Record Dates: First submitted 2024-11-25; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Voice Quality; Singing
Keywords: voice training; acoustic; respiratory therapy

STUDY DESIGN:
Intervention Model Description: all participants will perform adapted Lee Silverman Method (Adapt Lee) and Lung volume recruitment technique plus Adapt Lee during 2 weeks, with washout period of 6 weeks.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors will be blinded for intervention applied before the asessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adapted Lee Silverman Method (Active Comparator): The individuals will perform the Lee Silverman methods adapted to voice professionals. They will do a 14-day protocol, with three sets of 5 repetitions daily.
  Interventions: Procedure: Adapted Lee Silverman Method
- Lung volume recruitment Technique - LVRT (Experimental): In the LVRT intervention, the same exercises as in the adapted LEE Silverman intervention will be performed, however, a bag-mask ventilation system (Lumiar, Brazil) will be attached during the emission with an inflated oro-nasal mask (Lumiar, Brazil) connected to a pressure gauge (Illife device, Brazil) that will monitor the inspiratory pressure level between 30 and 40 cmH2O during phonatory emissions. it will be performed 3 sets with 5 repetitions.
  Interventions: Device: Lung volume recruitment technique - LVRT

INTERVENTIONS:
Procedure: Adapted Lee Silverman Method — Exercise protocol with 6 steps that the voice professionals adapted from Lee Silverman Method
  Arms: adapted Lee Silverman Method
Device: Lung volume recruitment technique - LVRT — The adapted Lee Silverman Method will have a addiction of LVRT technique. Lung inflation begins, reaching an optimal inspiratory peak of 30 cmH2O. From this point, the sound /HA/ begins to be emitted until the most comfortable low sound, where the emission should be maintained for as long as possible, making sure that this time is not less than 12 seconds, trying to emit a high and comfortable vocal intensity. When performing the emissions, the mouth should be kept wide open with the tongue, jaw and neck relaxed, repeating 5 emissions in 3 series. Between series, the participant will be instructed to drink 50 ml of water exactly as in the previous emissions.
  Arms: Lung volume recruitment Technique - LVRT

SUMMARY:
The goal of this clinical trial in voice professionals with both genders aimed to verify the changes in the vocal range profile and the changes in the glottic and vocal tract configuration for more efficient phonation after applying the adapted Lee Silverman Method and the addiction of lung volume recruitment technique in acoustic and structural analysis.

DETAILED DESCRIPTION:
A cross-over randomized trial with two arms-the Lee Silverman Method and the addiction of lung volume recruitment technique (LVRT)-will be conducted with voice professionals to assess the effects of both interventions on the acoustic, perceptive, and visual aspects of voice and their impact on respiratory muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Voice professionals with no voice disease

Exclusion Criteria:

* smokers
* Glottis paralysis and dysfunction
* dental problems
* Mental and cognitive disorders

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Vocal Range Profile | 30 days
  Minimum fundamental frequency - f0; Maximum f0; Extension f0; Extension in Semitone; Minimum intensity; Maximum intensity and Area

SECONDARY OUTCOMES:
functional laryngeal assessment | 30 days
  The Colton and Casper protocol will assess phonatory function using an endoscopic evaluation with a flexible fiberoptic endoscope.
Respiratory muscle strength | 30 days
  Dynamic inspiratory muscle strength (S-index) will be obtained using the KH5 device of the POWERbreathe®.

CONTACTS AND LOCATIONS:
Locations (1):
- Unievangelica, Anápolis, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No
a one center trial study without another institution linked with it